CLINICAL TRIAL: NCT01045122
Title: Sedation in Patients at Risk for Sleep-induced Upper Airway Collapse
Brief Title: Sedation in Patients at Risk for Upper Airway Collapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Suzanne Karan, Principal investigator, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Sleep Study CReFF award; 5M01RR000044 (NIH)
Record Dates: First submitted 2009-12-11; First posted 2010-01-08 (Estimated); Results first posted 2015-04-27 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Other): Is an alkylphenol, is primarily indicated for use as a general anesthetic and has minimal analgesic properties.
  Interventions: Drug: Propofol
- Dexmedetomidine (Other): Dexmedetomidine is an alpha-2 adrenoreceptor agonist that has sedative, hypnotic, and analgesic effects.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — For propofol, the current study will employ the Marsh parameters, with an initial effect site target concentration of 1.0 mcg/ml, a level likely to produce only mild sedation. Though our patient population is expected to be predominantly obese, a previous pharmacokinetic study has validated that constant infusions utilizing the dosing scheme of mcg-1•kg-1•min will yield similar effect site concentrations.25 The effect site target will be increased in increments approximately every five minutes until the pharmacodynamic targets defined in the study are attained.
  Other Names: Diprivan
  Arms: Propofol
Drug: Dexmedetomidine — For dexmedetomidine, an intravenous loading dose of 0.5 mcg/kg will be infused over 10 minutes and followed by an infusion starting at 0.5 mcg/kg/hr. This infusion will be titrated up to a maximum of 1.2 mcg/kg/hr.
  Other Names: Precedex
  Arms: Dexmedetomidine

SUMMARY:
Overview of Protocol:

Between Subject - Repeated Measures design will be used to assess the airway response of two groups of subjects under two different sedated conditions. Each group will be comprised of six subjects and will be categorized according to their baseline profile for risk for SDB (< 10 RDI or > 25 RDI). Some subjects will have been prescribed continuous positive airway pressure (CPAP) therapy by their treating physician as a result of their overnight sleep study. CPAP treatment is effective in splinting the airway open and thus decreasing the incident of airway collapse during sleep. Thus, CPAP utilization will also be tracked as an independent and continuous variable as regular CPAP use has been found to be associated with increased resistance to UAC (upper airway collapse).

The experimental conditions will evaluate upper airway patency and instability in response to two forms of intravenous sedation: propofol and dexmedetomidine.

Subjects will be continuously monitored during each experimental condition for respiratory effort and flow, and for EEG, EMG, and ECG.

Respiratory instability will first be assessed while subjects are under sedation without any airway provocation. The degree of respiratory instability will be quantified in terms of the following measurements: a modified Respiratory Disturbance Index (RDIsedated), respiratory arousals, and minute ventilation. The apneic periods will be classified by their mixture of central and obstructive components.All outcome measurements are assessed over the period of sedation which last for approximately one hour.

Upper airway patency will be quantified in terms of the critical pharyngeal pressure (Pcrit) (the pressure beyond which complete upper airway collapse occurs, see background).

DETAILED DESCRIPTION:
The propensity to experience sleep disordered-breathing (SDB) is controlled by the interplay of anatomic factors (i.e. BMI, neck circumference, retrognathia) and neurological drive (sleep stage, arousal). The interaction of baseline anatomic factors and drug-induced altered neurologic drive may also convey a risk for upper airway collapse (UAC) in patients receiving analgesics, or sedation/anesthesia.1;2 While there is mainly only anecdotal evidence to support the proposition that SDB is a strong predictor of sedation-related adverse events,3;4 there is such a remarkable consensus of opinion regarding this association that, for example, the American Society of Anesthesiologists is developing guidelines to specifically address the issue of managing this group of "at risk" patients who are to undergo sedation or anesthesia. SDB is a term that is used to describe a spectrum of sleep-related breathing disturbances. Obstructive Sleep Apnea (OSA) is a condition that incorporates SDB with daytime symptoms (i.e. hypersomnolence). These terms are commonly used interchangeably.

At this juncture, what is needed are clear demonstrations: 1) that SDB confers risk for sedation-related adverse events (epidemiologically and/or experimentally), 2) of the patient and drug factors that moderate/mediate the risk, and 3) of the mechanisms responsible for the patient by drug interactions.

This proposed project will, in a preliminary way, address the first and second of these issues. Specifically, the upper airway characteristics of patients with different severity classifications of SDB will be assessed while under the influence of two, neuropharmacologically distinct, intravenous sedatives.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild or no Sleep disorder breathing
* Patients with moderate to severe Sleep disorder breathing

Exclusion Criteria:

* No unstable medical conditions
* Anatomic pathology of airway
* Pregnancy or nursing
* Inability to fit an anesthesia facemask
* Excessive alcohol or drug abuse
* Bleeding abnormalities
* Claustrophobia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne B Karan, Medical, Principal Investigator — University of Rochester; Denham Ward, Medical, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment April 2006 to November 2008. Subjects were recruited from advertisements, patient letters sent out through the strong sleep center.
Pre-assignment Details: Subjects excluded from trial before assignment to group because Prior airway surgery, unstable medical conditions.
Groups:
- Propofol First: Propofol was administered first in 5/11 subjects with a one week washout at least between the next run with dexmedetomidine
- Dexmedetomidine First: Dexmedetomidine was administered on the first day in 6/11 subjects with at least a one week washout between runs before the subjects underwent the experiment with propofol.
Period: Dexmedetomidine Then Propofol
Arm/Group | Propofol First | Dexmedetomidine First
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Propofol Then Dexmedetomidine
Arm/Group | Propofol First | Dexmedetomidine First
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Propofol vs Dexmedetomidine: We aim to study two commonly used sedatives (propofol vs dexmedetomidine) in subjects with OSA for their propensity to produce sedation related respiratory events
Arm/Group | Propofol vs Dexmedetomidine
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 11
Respiratory Disturbance Index [Mean (Standard Deviation); unit: events per hour] — The Degree of respiratory instability will be quantified in terms of the following measurements: a Respiratory Disturbance Index in events per hour.
  events per hour | 39.99 (40.1)

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Disturbance Index
Description: respiratory events (apneas, hypopneas) per hour
Time Frame: during infusion of study drugs
Population: Per protocol
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- Propofol; Dexmedetomidine: The respiratory disturbance index and airway closing pressures (Pcrit) were quantified for both arms
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 11 | 11
events per hour | 57.52 (165.6) | 21.32 (39.2)

ADVERSE EVENTS:
Arm/Group | Propofol | Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes